CLINICAL TRIAL: NCT04244396
Title: Persistent AF (Asia Pacific) Observational Study
Brief Title: Persistent Atrial Fibrillation (AF) APAC (Asia Pacific) Observational Study
Acronym: PerAF APAC
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early by the Sponsor as sufficient data had been collected to satisfy the study objectives.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10295
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Radiofrequency Ablation; Heart Disease; Tachycardia; Cardiovascular Diseases; Cardiac Conduction System Disease; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Heart Diseases; Tachycardia; Cardiovascular Diseases; Cardiac Conduction System Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Drug refractory, symptomatic persistent atrial fibrillation: Asian population
  Interventions: Device: TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE)

INTERVENTIONS:
Device: TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE) — TactiCath SE is indicated for use in cardiac electrophysiological mapping (stimulation and recording), and, when used in conjunction with a radiofrequency generator, for cardiac ablation of supraventricular arrhythmias in the right and left atrium, including atrial fibrillation.

SUMMARY:
The objective of this clinical trial is to collect safety and effectiveness data for the TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE) in the APAC patient population for the treatment of drug refractory, symptomatic persistent atrial fibrillation when following standard electrophysiology mapping and radiofrequency (RF) ablation procedures.

DETAILED DESCRIPTION:
The PerAF APAC trial is a prospective, single arm, non-randomized, observational, post-market clinical investigation. Approximately 100 subjects will be enrolled at up to 15 sites in South Korea, Singapore, Hong Kong, Taiwan, and India. Centers in other countries within APAC may be approached for participation in the clinical investigation as needed. Subjects will be followed for 15-months after their initial ablation procedure. The primary effectiveness and safety endpoints will be evaluated through 15-months. A core lab will independently assess AF/Atrial Flutter (AFL)/(Atrial tachycardia (AT) recurrence via Holter monitoring at the 6-month and 15-month follow-up visits. All serious adverse events (SAEs) will be independently adjudicated by qualified physicians not participating in the trial

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Documented symptomatic persistent AF, defined as continuous AF sustained >7-days but <1 year documented by:

   1. Physician's note AND one of the following:
   2. 24-hr Holter showing continuous AF within 90-days of the procedure OR
   3. 2 ECGs (from any form of rhythm monitoring) showing continuous AF, taken at least 7-days apart
3. Refractory or intolerant to at least one Class I or III antiarrhythmic drug (AAD) as evidenced by recurrent symptomatic AF Note: Intolerant = unable, unwilling, or refusal to take AADs
4. ≥18 years of age
5. Able and willing to complete all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

1. Continuous AF >12 months (longstanding persistent AF)
2. Previous left atrial (LA) surgical or catheter ablation for AF
3. Any cardiac procedure within 90-days prior to initial procedure (Diagnostic procedures with no intervention are not considered a surgical or percutaneous surgical procedure)
4. Coronary artery bypass graft (CABG) surgery within 6-months (180-days) prior to initial procedure
5. Valvular cardiac surgical/percutaneous procedure (i.e. ventriculotomy, valve repair or replacement and/or presence of a prosthetic or mechanical valve)
6. Any carotid stenting or endarterectomy
7. Documented or known left atrial thrombus on imaging
8. Left atrial (LA) diameter >50 mm (parasternal long axis view or by CT)
9. Left Ventricular Ejection Fraction (LVEF) <40%
10. Unable to take anticoagulation medication due to contraindication or intolerance
11. History of blood clotting or bleeding abnormalities
12. Myocardial Infarction (MI), acute coronary syndrome, Percutaneous coronary intervention (PCI) within the 3-months (90-days) prior to the initial procedure
13. Documented thromboembolic event (including TIA) within 12-months (365 days) prior to the initial procedure
14. Rheumatic heart disease
15. Uncontrolled heart failure or New York Heart Association (NYHA) Class III or IV
16. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2)
17. Awaiting cardiac transplantation or other cardiac surgery within 12-months (365 days) following the initial ablation procedure
18. Unstable angina at the time of the initial procedure
19. Acute illness or active systemic infection or sepsis
20. AF secondary to electrolyte imbalance, thyroid disease, acute alcohol intoxication, major surgical procedure in the preceding 3-months, or other reversible or non-cardiac cause
21. Diagnosed atrial myxoma
22. Presence of implanted implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy-defibrillator (CRT-D)
23. Significant pulmonary disease, (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
24. Significant congenital anomaly or other anatomic or comorbid medical problem that in the opinion of the investigator would preclude enrollment in this study or compliance with the follow-up requirements or impact the scientific soundness of the clinical trial results
25. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period
26. Enrollment in an investigational study evaluating another device, biologic, or drug that may interfere with this clinical investigation at the time of the initial procedure or within 30 days prior to the initial procedure
27. Presence of any condition that precludes appropriate vascular access or manipulation of catheter
28. Life expectancy less than 12-months
29. Body mass index >40 kg/m2
30. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
31. Renal failure requiring dialysis
32. Presence of other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results
33. History of atriotomy or ventriotomy
34. Implanted left atrial appendage occlusion device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll drug refractory, symptomatic, persistent atrial fibrillation (AF) subjects who will undergo a de novo RF ablation procedure. Subjects must provide written informed consent prior to conducting any investigation-specific procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, Study Director — Abbott
Locations (9):
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Singapore (2):
  - National Heart Centre Singapore, Singapore
  - National University Hospital, Singapore
- South Korea (3):
  - Sejong Hospital, Bucheon-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Centre, Soeul
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
- Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug Refractory, Symptomatic Persistent Atrial Fibrillation
Started | 82
Procedure Completed | 81
7-Day Follow-up | 81
14-Day Follow-up | 81
3-Month Follow-up | 79
6-Month Follow-up (Withdraw prior to 6M visit N = 4) | 76
12-Month Follow-up (Withdraw prior to 12M visit N = 22) | 54
15-Month Follow-up (Withdraw prior to 15M visit N = 13) | 37
Completed | 42
Not Completed | 40
Not completed — Subject did not meet screening inclusion/exclusion criteria | 1
Not completed — Withdrawal by Subject | 2
Not completed — Study termination | 37

BASELINE CHARACTERISTICS:
Arm/Group | Drug Refractory, Symptomatic Persistent Atrial Fibrillation
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 81
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 38
  Singapore | 12
  Hong Kong | 6
  Taiwan | 18
  Thailand | 7

OUTCOME MEASURES:

1. Primary Outcome: Rate of Device and/or Procedure-related Serious Adverse Events
Description: device and/or procedure-related serious adverse events are pre-defined as below with onset within 7-days of any ablation procedure that uses the TactiCath SE catheter (initial or repeat procedure performed ≤180 days of initial procedure)
  * Atrioesophageal fistula - assessed through 15 months
  * Cardiac tamponade/perforation - assessed through 15 months
  * Death
  * Heart block
  * Myocardial infarction (MI)
  * Pericarditis - pleuritic symptoms >7 days and/or requires hospitalization >24 hrs for reasons other than observational purposes only
  * Phrenic nerve injury resulting in diaphragmatic paralysis
  * Pneumothorax
  * Pulmonary edema (respiratory insufficiency)
  * Pulmonary vein stenosis - assessed through 15 months
  * Stroke/cerebrovascular accident
  * Thromboembolism
  * Transient ischemic attack
  * Vascular access complications (including major bleeding events)
Time Frame: Through 7-days
Population: The primary safety endpoint was the rate of pre-specified device and/or procedure-related serious adverse events with onset within 7-days of any ablation procedure that used the TactiCath SE catheter (initial or repeat procedure performed ≤180 days of initial procedure), with the exception of atrio-esophageal fistula, cardiac tamponade/perforation, and pulmonary vein stenosis which were evaluated through 15-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Refractory, Symptomatic Persistent Atrial Fibrillation
Number analyzed (Participants) | 81
Participants | 3

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Drug Refractory, Symptomatic Persistent Atrial Fibrillation
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 16/81
Other Adverse Events (participants affected / at risk) | 3/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Refractory, Symptomatic Persistent Atrial Fibrillation (N=81)
Arrhythmia (Cardiac disorders) | 2 (2)
Bleeding/Anemia (Blood and lymphatic system disorders) | 2 (2)
Cerebrovascular Accident/ Stroke (Blood and lymphatic system disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Volume Overload (Blood and lymphatic system disorders) | 1 (1)
Chest Pain/Discomfort (Cardiac disorders) | 1 (1)
Elective Procedure/Surgery (General disorders) | 1 (1)
Heart Failure/Pump Failure (Cardiac disorders) | 2 (3)
Acute Gout (General disorders) | 1 (1)
Common Bile Duct Stone With Cholangitis (General disorders) | 1 (1)
Finger Fracture (General disorders) | 1 (1)
Unexplained Jaundice And Raised Liver Panel (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Refractory, Symptomatic Persistent Atrial Fibrillation (N=81)
Arrhythmia (Cardiac disorders) | 1 (1)
Vascular Bleeding/Local Hematomas/Ecchymosis (Blood and lymphatic system disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
In April 2022, communication was sent to sites informing them that enrollment was ending. The number of subjects enrolled at the time was deemed sufficient to assess the study endpoints while maintaining the study completion timelines. Follow-up was to continue as scheduled for those already enrolled and those enrolled prior to the end enrollment date of 30 April 2022. In September 2022, sufficient data had been collected so a decision was made to fully close the PerAF APAC clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The data and results from the clinical investigation are the sole property of the Sponsor. The Investigators will not use this clinical investigation-related data without the written consent of the Sponsor for any purpose other than for clinical investigation completion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04244396/Prot_SAP_000.pdf